CLINICAL TRIAL: NCT07376967
Title: Improving Healthcare Outcomes With Early Detection of Liver Related Complications in Liver Cirrhosis Patients by Implementing a Telemedicine Care Pathway (myLIVERcoach): a Multicenter Feasibility Study
Brief Title: Improving Healthcare Outcomes With Early Detection of Liver Related Complications in Liver Cirrhosis Patients by Implementing a Telemedicine Care Pathway (myLIVERcoach)
Acronym: myLiverCOACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Dutch Digestive Diseases Foundation (Other); Gelre Hospitals (Other); Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: METC 2022-3567
Record Dates: First submitted 2023-05-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Liver Cirrhosis
Keywords: Telemedicine; eHealth; Telemonitoring; mobile health
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using telemedicine on top of standard care (Other)
  Interventions: Device: telemedicine pathway

INTERVENTIONS:
Device: telemedicine pathway — Patients are able to use an online application on top of standard care. Monitoring complications, subjective wellbeing and lifestyle factors. Patients are able to go through information about liver cirrhosis and additional aspects, like dietary advices, at any moment in time. Furthermore, they are able to contact their healthcare professional through the chat function.

SUMMARY:
The goal of this multicenter feasibility study is to investigate the feasibility of our telemedicine platform (myLIVERcoach) in liver cirrhosis patients, according to liver cirrhosis patients, caregivers and healthcare professionals. The main question[s] it aims to answer are:

1. What is the feasibility of a telemonitoring pathway according to patients, caregivers and healthcare professionals in liver cirrhosis care?

   Secondary objectives:
2. What is the level of acceptability, usability, learnability and desirability of a telemonitoring pathway in liver cirrhosis care from the patients, caregivers and healthcare professionals' perspective?
3. What is the level of compliance of patients, caregivers and healthcare professionals using a telemonitoring pathway in liver cirrhosis care?
4. What is the occurrence of liver related complications in liver cirrhosis patients using a telemonitoring pathway?
5. What is the occurrence of clinical admissions and emergency concultations in liver cirrhosis patients using a telemonitoring pathway?
6. What is the mortality rate in liver cirrhosis patients using a telemonitoring pathway?

8. What is the effect of a telemonitoring pathway on patients perceived health, quality of life and work participation of liver cirrhosis patients?

Participants will be asked to use myLIVERcoach on top of standard care. According to disease stadium participants will receive different online questionnaires and measurements, focusing on early detection of complications and psychosocial and lifestyle factors. Participants are able to contact their healthcare professional and go through information about their disease as well.

After six months, participants will be asked to fill out a questionnaire regarding their experiences with myLIVERcoach in order to optimize the system. In addition the investigators will perform interviews with ten patients or caregivers and with healthcare professionals at the end of follow-up.

DETAILED DESCRIPTION:
Methods Study parameters/endpoints Main study parameter/endpoint Feasibility of this telemonitoring pathway in liver cirrhosis patients will be defined by results of the acceptability questionnaire, appendix B.

A score of ≥4.0 in ≥70% of patients, caregivers and healthcare professionals together will be defined as feasible.

Results of the question ''I would recommend the application to others'', see appendix B. A score ≥4.0 in ≥70% of patients, caregivers and healthcare professionals together is defined as significant satisfaction, one of the main aspects of adequate feasibility.

Feasibility will be evaluated in the interviews as well. The telemonitoring pathway will be defined feasible if ≥70% of interviewed patients and at least three (out of five) healthcare professionals find the telemonitoring of value in the domains: acceptance of implementation in standard liver cirrhosis care, support of self-management and adequate technological functioning.

Secondary study parameters

1. Compliance is divided into responsiveness to questionnaires and e-learnings and completion of questionnaires and e-learnings.

   1. Adequate compliance regarding responsiveness is defined as ≥70% of patients and caregivers starting the provided questionnaires and e-learnings.
   2. Adequate compliance regarding completion is defined as ≥70% of patients and caregivers completing the provided questionnaires and e-learnings.
2. Usability, learnability, and desirability are defined as a mean score of ≥4.0 in ≥70% patients, caregivers, and healthcare professionals together.
3. Occurrence of liver related complications (ascites, hepatic encephalopathy, and variceal bleeding) will be described using percentage of occurred complication and how many times patients developed this complication.
4. Occurrence of clinical admissions will be described using percentage of occurred clinical admissions and how often patients were admitted.
5. Emergency consultations will be described using percentage of occurred emergency consultation and how many times patients had those consultations.
6. Mortality will be described using percentage of occurred death.
7. Perceived health will be monitored before and after follow-up and the investigators will investigate significant differences in disease status within patients before and after using the telemonitoring pathway.
8. Quality of life will be monitored before and after follow-up and the investigators will investigate significant differences in quality of life within patients before and after using the telemonitoring pathway.
9. Work participation will be monitored before and after follow-up and the investigators will investigate significant differences in work participation within patients before and after using the telemonitoring pathway.
10. Social functioning will be monitored before and after follow-up and the investigators will investigate significant differences in social functioning within patients before and after using the telemonitoring pathway.
11. Adequate detection of complications will be classified as ≥70% of complication specific exceeding thresholds in myLIVERcoach leading to change in treatment
12. Adequate comprehensibility of the liver complication specific questionnaire according to patients, caregivers and healthcare professionals will be classified as ≥70% acknowledgement during the interviews of understanding all the individual questions.

Data collection Research data from myLIVERcoach will be coded, encrypted, and stored in repositories of Datahub Maastricht, a so called trusted third party. Data conducted from the electronic patient files will be stored in Castor. Every participating hospital will manage research data of their specific patients. Key documents, to which just the principal investigator and coordinating researcher have access, will be saved separately in the participating hospitals.

Patients and caregivers During a study period of 6 months, patients will fill in questionnaires in myLIVERcoach regarding disease specific complaints, quality of life and subjective wellbeing in intervals according to the group participants are subjected to (compensated, non-actively decompensated and actively decompensated). Participants will complete separate questionnaires regarding satisfaction with current healthcare and acceptability of the telemonitoring pathway at baseline and at 6 months. Caregivers will fill in questionnaires regarding current healthcare for the patient and will be asked to complete the myLIVERcoach questionnaires together with the patient. The investigators will evaluate different aspects with ten to twenty patients using the telemonitoring pathway in a semi-structured 30-60-minute interview.

The investigators can measure patients and caregivers' compliance to the modules and questionnaires of the telemonitoring pathway in terms of starting a module, completing it and duration until completion. The investigators will search electronic patient files to investigate occurrence of liver related complications, clinical admissions, emergency consultations and mortality.

Healthcare professionals During 6 months, healthcare professionals are able to monitor patients' responses to questions and e-learnings and receive alarm signals in case of exceeding thresholds. Participants will complete separate questionnaires regarding satisfaction acceptability of the telemonitoring pathway at baseline and at 6 months. The investigators will evaluate different aspects including compliance with at least 5 healthcare professionals in a semi-structured 30-60-minute interview.

Design and content development The backbone of the technical system and general content of our telemonitoring system is based on myIBDcoach. This is a well-tested and validated digital platform that supports the healthcare provider in monitoring, guiding, educating, and communicating with patients diagnosed with inflammatory bowel diseases (IBD) [17]. The investigators were able to use approximately 60% of the general content in myIBDcoach. Decisions regarding which general and liver-specific content should be included in our telemonitoring pathway were made in brainstorm sessions of our content committee. The content committee included a representative from the Dutch Liver Patient Association (NLV), a hospital pharmacist, 4 gastroenterologists/hepatologists (academic/non-academic and including an electronic Health expert), a dietician, 2 specialized hepatology nurses, a physical therapist and a clinical researcher who is responsible for continuation, development and contact with the software provider. In the 2 months prior to start of the feasibility study our content committee has iteratively tested and reviewed our telemonitoring pathway after which it has been improved and tested again until it was found worthy for patient use in the feasibility study. See fig. 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age or caregiver of a patient (both ≥ 18 years of age)
* Liver cirrhosis, based on biopsy, fibroscan or diagnostic imaging data or caregiver of a patient with this diagnosis

Exclusion Criteria:

* Inability to read or understand informed consent
* Lack of internet access
* History of or current hepatocellular carcinoma
* History of or current hepatic metastasis
* History of liver transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Feasibility defined by the number of recommendations to use this telemonitoring pathway by patients, caregivers and healthcare profesionals. | 6 months
  A score of ≥4.0 in ≥70% of patients, caregivers and healthcare professionals together will be defined as feasible.
  Using a likert scale, minimum value 1 (worst), maximum value 5 (best) Results of the question ''I would recommend the application to others'', see appendix B. A score ≥4.0 in ≥70% of patients, caregivers and healthcare professionals together is defined as significant satisfaction, one of the main aspects of adequate feasibility.

SECONDARY OUTCOMES:
Compliance defined by ≥70% initiated questionnaires and e-learnings of actual provided questionnaires and e-learnings. | 6 months
  Using a percentage based upond the number of provided questionnaires and the number of questionnaires actually initiated by patients and caregivers.
Compliance defined by ≥70% completed questionnaires and e-learnings of actual provided questionnaires and e-learnings. | 6 months
  Using a percentage based upond the number of provided questionnaires and the number of questionnaires actually completely finished by patients and caregivers.
Usability defined as a mean score of ≥4.0 in ≥70% patients, caregivers, and healthcare professionals together in the question ''It was easy to indicate my complaints with myLIVERcoach.'' | 6 months
  Using a likert scale, minimum value 1 (worst), maximum value 5 (best)
Learnability defined as a mean score of ≥4.0 in ≥70% patients, caregivers, and healthcare professionals together in the question ''It was easy to learn how I had to use myLIVERcoach''. | 6 months
  Using a likert scale, minimum value 1 (worst), maximum value 5 (best)
Desirability defined as a mean score of ≥4.0 in ≥70% patients, caregivers, and healthcare professionals togethe in the question ''MyLIVERcoach meets my approval.'' | 6 months
  Using a likert scale, minimum value 1 (worst), maximum value 5 (best)
Number of liver related complications | 6 months
Clinical admissions | 6 months
  Occurrence of clinical admissions will be described using percentage of occurred clinical admissions and how often patients were admitted.
Emergency consultations | 6 months
  Emergency consultations will be described using percentage of occurred emergency consultation and how many times patients had those consultations.
Mortaility | 6 months
  Mortality will be described using percentage of occurred death.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Gelre Ziekenhuizen, Apeldoorn, Gelderland
  - Maastricht University Medical Center, Maastricht, Limburg

IPD SHARING:
Plan to Share IPD: No